CLINICAL TRIAL: NCT01521845
Title: Phase 3 Study of Poly Unsaturated Fatty Acids of Omega 3 as an Anti Platelet Agent on Biomarkers of Cardiac Necrosis Including CKMB and Troponin I and Inflammation Marker CRP
Brief Title: Study of the Effect of omega3 on Biomarkers of Cardiac Necrosis (CKMB and Troponin I) and Inflammation Marker (CRP) After Elective Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jamshid Salamzadeh, PhD, PhD, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90-1-94-8048
Record Dates: First submitted 2012-01-19; First posted 2012-01-31 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Arteriosclerosis
Keywords: elective percutaneous coronary intervention; hs-CRP; CKMB and troponin I
MeSH Terms: conditions — Coronary Artery Disease | interventions — Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- omega 3 (Active Comparator): receive omega 3 in addition to standard treatment
  Interventions: Drug: omega 3
- control (No Intervention): This group is without omega 3 : just receives standard treatment

INTERVENTIONS:
Drug: omega 3 — 3 gram omega 3 (400mg EPA and 200mg DHA) 12hours before PCI
  Other Names: fish oil
  Arms: omega 3

SUMMARY:
The purpose of this study is to investigate the effect of omega 3 on biomarkers of cardiac necrosis(CKMB and troponin I) and inflammation marker CRP.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) has become the most common form of coronary revascularization worldwide. Although PCI is a safe procedure, it may have multiple risks including bleeding, coronary dissection, abrupt vessel closure, and myocardial necrosis. It is estimated that approximately 25% of patients undergoing PCI have significant postprocedural creatinine kinase (CK)/creatinine kinase myocardial band (CK-MB) elevations and approximately 50% of patients have significant post-procedural troponin elevations. Initially, it was felt these elevations were simple enzyme leaks with no long-term implications.

Now, several studies have demonstrated that periprocedural infarction is associated with short-, intermediate-, and long-term adverse outcomes, most notably mortality. Pretreatment with antiplatelets such as aspirin and clopidogrel play an important role in reducing cardiovascular events (CV events) following PCI.

Omega -3 polyunsaturated fatty acids (PUFAs) have antiplatelet effect. It may also improve response to aspirin and clopidogrel in low-response patients.

This study is a randomized clinical trial (RCT) evaluating the effect of omega 3 supplement [with 400mg Eicosapentaenoic acid (EPA) and 200mg docosahexanoic acid (DHA)] on biomarkers of cardiac necrosis (CKMB and troponin I) in patients undergoing elective PCI. Eighty patients planed to do elective PCI will be categorized into two groups. The first group will be received standard regimen for PCI (aspirin, clopidogrel, and heparin) and the second group will be treated with standard regimen in addition to 3 gram omega 3 (12 hours before PCI). Blood samples will be drawn in all patients before and 8 and 24 h after intervention for cardiac biomarkers assessment (CK-MB, troponin I)and inflammation marker C-reactive protein (CRP). Major adverse cardiac events (MACE) will be evaluated as a second endpoint.

ELIGIBILITY:
Inclusion Criteria:

* candidate of elective PCI
* treatment with aspirin at least 5 days before PCI

Exclusion Criteria:

* high CKMB and troponin I level
* cardiac bypass in recent 3 months
* platelet count < 70×10 9/L
* sever chronic renal failure
* active bleeding
* treatment with glycoprotein IIb/IIIa inhibitors during PCI
* treatment with bivalirudin during PCI
* sensitivity to aspirin and clopidogrel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Salamzadeh, PhD, Principal Investigator — SBMU School of Pharmacy; farzaneh foroughinia, phD, Study Director — Shiraz University of Medical Sciences
Locations (1):
- Moddaress Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Foroughinia F, Salamzadeh J, Namazi MH. Protection from procedural myocardial injury by omega-3 polyunsaturated fatty acids (PUFAs): is related with lower levels of creatine kinase-MB (CK-MB) and troponin I? Cardiovasc Ther. 2013 Oct;31(5):268-73. doi: 10.1111/1755-5922.12016. PMID 23134549

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega 3 | Control
Started | 52 | 52
Completed | 43 | 47
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega 3 | Control | Total
Number analyzed (Participants) | 43 | 47 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 60 (11) | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 27 | 33 | 60
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 43 | 47 | 90

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Necrosis Biomarkers (CKMB, Troponin I)
Description: difference between study and control group in 8 and 24 hrs after percutaneous coronary intervention
Time Frame: 8 and 24 hrs after percutaneous coronary intervention
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Omega 3 | Control
Number analyzed (Participants) | 43 | 47
ng/ml | 13 [10 to 18] | 18 [13 to 23]
Statistical Analysis 1: Comparison: Omega 3 vs Control; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Inflammation Marker (CRP)
Description: difference between study and control group in 8 and 24 hrs after percutaneous coronary intervention
Time Frame: 8 and 24 hrs after percutaneous coronary intervention
Measure: Median (Inter-Quartile Range); unit: mg/l
Arm/Group | Omega 3 | Control
Number analyzed (Participants) | 43 | 47
mg/l | 3 [1 to 10] | 6 [2 to 15]
Statistical Analysis 1: Comparison: Omega 3 vs Control; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: MACE(Major Adverse Cardiac Effect) Defined as Need for Target Revascularization, Myocardial Infarction and Death
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Omega 3 | Control
Number analyzed (Participants) | 43 | 47
participants | 0 | 0
Statistical Analysis 1: Comparison: Omega 3 vs Control; Test type: Superiority or Other; p = 1, not comparable

ADVERSE EVENTS:
Arm/Group | Omega 3 | Control
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/47
Other Adverse Events (participants affected / at risk) | 0/43 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes